CLINICAL TRIAL: NCT04805021
Title: Acquired Hemophilia A and Autoimmunity. Study of Lymphocyte Populations and Myeloid-Derived Suppressor Cells
Acronym: IMMUNHEMAC
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0253
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — a tube of blood taken from CTAD or citrate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients in the Acquired Hemophilia A group.
  Interventions: Other: no intervention
- patients in the constitutional hemophilia A group.
  Interventions: Other: no intervention
- patients in the control subjects group.
  Interventions: Other: no intervention
- patients in the group of patients with inflammatory pathology.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Acquired hemophilia A is a rare condition of hemostasis secondary to the development of antibodies against factor VIII. This is a potentially serious pathology that can be life-threatening due to the major risk of bleeding caused by the sometimes drastic decrease in the level of circulating factor VIII.

This pathology occurs overwhelmingly in elderly subjects or, more rarely, in young women, during the postpartum period. It appears idiopathic in 50% of cases and associated, for the other cases, with underlying pathologies such as autoimmune pathologies (rheumatoid arthritis and bullous pemphigoid in particular) and neoplasias, or with a particular circumstance represented by the post -partum.

The association between this autoimmune pathology and its association with pathologies of the same type or with circumstances involving the immune system, suggests that common mechanisms could favor its emergence.

This study therefore proposes to study lymphocyte populations and subpopulations as well as Myeloid-Derived Suppressor Cells and the cytokine profile, which are abnormal in a large part of autoimmune pathologies.

ELIGIBILITY:
Inclusion Criteria:

1. Patient population with acquired hemophilia A:

   Adult patients with a diagnosis of acquired hemophilia A and with a social security system. Obtaining oral non-opposition from the patient to participate in the study following the submission of an information note relating to the project.

   Obtaining signed and written informed consent for biocollection consent.
2. Population of Patients with constitutional hemophilia A:

   Adult patients over 50 years of age with severe or moderate constitutional hemophilia A, with no history of autoimmune disease, and with a social security system.

   Obtaining oral non-opposition from the patient to participate in the study following the submission of an information note relating to the project.

   Obtaining signed and written informed consent for biocollection consent.
3. Population of control subjects:

   Adult patients, over the age of 60, without a coagulation abnormality, with no history of autoimmune disease, and with a social security system.

   Obtaining oral non-opposition from the patient to participate in the study following the submission of an information note relating to the project.

   Obtaining signed and written informed consent for biocollection consent.
4. Patient population with inflammatory pathology:

Adult patients over the age of 50 with an inflammatory pathology likely to be associated with acquired hemophilia A, and with a social security system.

Obtaining oral non-opposition from the patient to participate in the study following the submission of an information note relating to the project.

Obtaining signed and written informed consent for biocollection consent.

Exclusion Criteria:

For the 4 groups:

* Minor patient, under guardianship or curatorship.
* Pregnant and lactating women.
* Blood transfusion less than 7 days old.
* Treatment with corticosteroids in the 7 days preceding inclusion or any other immunomodulatory or immunosuppressive treatment in the 4 weeks preceding inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acquired hemophilia A will be recruited prospectively when diagnosed with acquired hemophilia A and will be followed in the study until recovery.
  Patients with constitutional hemophilia A will be recruited prospectively. They should be over 50 years old and have severe or moderate hemophilia A, and not be taking any treatment that could interfere with the immune system or inflammatory markers.
  Population of control subjects without coagulation abnormalities, over 60 years of age and not taking any treatment likely to interfere with the immune system or inflammatory markers.
  Patient population with inflammatory pathology will include subjects with an inflammatory pathology likely, according to the literature, to be associated with acquired hemophilia A and, in particular patients with rheumatoid arthritis, if possible at diagnosis and not taking any treatment likely to interfere with the disease. immune system or inflammatory markers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the evolution of lymphocyte populations and subpopulations, MDSCs and inflammatory cytokines in patients with hemophilia A acquired at diagnosis and during follow-up | 2 years
  Comparisons between diagnosis and during follow-up

SECONDARY OUTCOMES:
To test the link between the severity of the disease at diagnosis and the cellular and cytokine parameters. | 2 years
  Factor VIII level and inhibitor titration at diagnosis
Comparisons of baseline lymphocyte and cytokine data between patients with a favorable versus unfavorable final diagnosis. | 2 years
  Cell populations and cytokine profile and half-life of the inhibitor under treatment, time before normalization of the Factor VIII / Willebrand factor ratio, total duration of treatment with corticosteroids, recurrence and mortality tested to define a favorable course of the disease or unfavorable.
Comparison of lymphocyte populations and subpopulations, MDSCs and inflammatory cytokines between different groups. | 2 years
  Cell populations and cytokine profile of the different groups at diagnosis and at the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fouassier, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - CHU de Nantes, Nantes
  - CH de Saint Nazaire, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: Undecided